CLINICAL TRIAL: NCT06371794
Title: Exploring Novel Molecular Determinants of Dravet Syndrome Phenotype Heterogeneity
Acronym: EXEDRA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: IRCCS San Raffaele (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ID 5460
Record Dates: First submitted 2024-04-03; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Dravet Syndrome
MeSH Terms: conditions — Epilepsies, Myoclonic

STUDY DESIGN:
Intervention Model Description: The ethics committee of the foundation FPG considers the study interventional since patients will undergo skin biopsy procedures ( around 4 mm)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- To characterize in detail and classify the DS phenotype (Other): Patients will be stratified according to the severity of epilepsy and cognitive impairment as follows:
  i) Severely impaired with severe epilepsy (SISE); ii) Severely impaired with mild epilepsy (SIME); iii) Mildly impaired with severe epilepsy (MISE); iv) Mildly impaired with mild epilepsy (MIME). Mild epilepsy will be defined by: i) no history of myoclonic and/or absence seizure; ii) no history of status epilepticus; iii) seizure frequency less than weekly. Patients not fulfilling these criteria will be considered as having severe epilepsy. Cut-off for severe impairment will be defined as a z-score of more or less of -3 of adaptive behavioral or intellectual abilities scales (vineland, WISC or equivalent).
  Interventions: Procedure: skin punch biopsy

INTERVENTIONS:
Procedure: skin punch biopsy — skin punch biopsy (around 4 mm2) from each studied subject.

SUMMARY:
Dravet syndrome is characterized as a developmental encephalopathy resulting from mutations of SCN1A, the gene encoding the alpha subunit of the voltage-gated sodium channel Nav1.1. The syndrome typically presents with drug-resistant epilepsy and varying degrees of cognitive disorders. Current treatment efficacy may be hindered by insufficient knowledge of undiscovered molecular determinants of the disease and its heterogeneous nature. Utilizing induced pluripotent stem cells (iPSCs) derived from skin biopsies, accessibility to patients' brain neurons has enabled successful modeling of various genetic neurological diseases. Neurons and brain organoids will be obtained from Dravet syndrome patients exhibiting diverse phenotypic severities, encompassing behavioral and developmental delays, to discern the molecular determinants of phenotypic diversity. Specifically, emphasis will be placed on investigating cellular and molecular mechanisms linking altered neuronal excitability with synaptic dysfunction.The study will focus on exploring the expression of newly identified modifiers potentially associated with neuronal excitability and synaptic function in iPSC-derived human neurons. This aims to establish correlations between the severity of epileptic and cognitive phenotypes and the altered expression of these proteins, whose functions are not fully understood.In the mid to long term, efforts will be directed towards overcoming the limitations of conventional therapeutic approaches for Dravet syndrome. This will involve attempting to reverse the observed morphological and functional alterations in Dravet syndrome neurons using viral vectors to promote overexpression/downregulation of identified modifiers correlated with disease severity. The anticipated outcomes of this project are expected to unveil novel molecular mechanisms underlying the pathophysiology of this severe neurogenetic disease, characterized by varying degrees of cognitive impairment. Moreover, these findings may pave the way for the discovery of innovative therapeutic strategies.

DETAILED DESCRIPTION:
Dravet Syndrome (DS) is characterized as both an epileptic encephalopathy, where seizures contribute to phenotype severity, and a developmental encephalopathy, where genetic background directly impacts developmental delay independently from seizure activity. The syndrome exhibits significant heterogeneity in phenotype severity, with polymorphic seizures typically occurring before age 12 months and progressing with varying severity. Additionally, cognitive and behavioral impairments become apparent during the second year of life or later, worsening with age and seizure frequency. Factors limiting the efficacy of current treatments likely include insufficient knowledge of unknown molecular determinants of the disease and its heterogeneity. To address this, novel molecular modifiers linked to excitability and synaptic function are hypothesized to unveil the pathophysiology of DS phenotype heterogeneity. The study aims to investigate hiPSCs-derived neurons from DS patients compared with age-matched healthy subjects. Specifically, skin biopsies will be obtained from DS patients and healthy controls to generate neurons and brain organoids. These models will be utilized to understand how changes in excitability and synaptic function affect phenotype severity in DS and to identify new molecular determinants associated with altered neuronal excitability and synaptic dysfunction. Aims of the study include classifying the epileptic and cognitive/behavioral phenotype severity of DS patients, characterizing neurons and brain organoids obtained from DS patients, and identifying potential phenotype modifiers. Additionally, the study aims to provide proof of concept for the development of novel modifier-related pharmacogenetic strategies to alleviate or rescue DS phenotype. Recruitment of DS patients and healthy controls will be conducted, and various assessments will be performed to classify phenotype severity. Functional, morphological, and molecular alterations in human neurons derived from DS patients will be investigated using a range of experimental techniques. Ultimately, the study seeks to deepen understanding of DS pathophysiology, identify potential therapeutic targets, and pave the way for personalized medicine approaches tailored to individual patients' molecular profiles.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed clinical diagnosis of Dravet Syndrome;
* Identification of a pathogenic variant in the SCN1A gene;
* Age between 18 and 35 years.

Exclusion Criteria:

- The presence of a significant neurological condition unrelated to Dravet Syndrome.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
TO CLASSIFY THE COGNITIVE/BEHAVIORAL PHENOTYPE SEVERITY OF DS PATIENTS | Through study completion, an average of 2 years
  Neuropsychological assessment of cognitive evaluation (Wechsler Adult Intelligence Scale)

SECONDARY OUTCOMES:
TO CLASSIFY THE COGNITIVE/BEHAVIORAL PHENOTYPE SEVERITY OF DS PATIENTS | Through study completion, an average of 2 years
  Neuropsychological assessment of adaptive behavior (Vineland-II scale).

OTHER OUTCOMES:
TO CLASSIFY THE COGNITIVE/BEHAVIORAL PHENOTYPE SEVERITY OF DS | Through study completion, an average of 2 years
  Neuropsychological assessment of psychiatric issues (Aberrant Behaviour Checklist)
TO CLASSIFY THE BEHAVIORAL PHENOTYPE SEVERITY OF DS PATIENTS | Through study completion, an average of 2 years
  Electrophysiological assessment: wake and sleep video-EEG and EMG monitoring
TO CLASSIFY THE BEHAVIORAL PHENOTYPE SEVERITY OF DS PATIENTS | Through study completion, an average of 2 years
  Motor assessment: characterization of movement disorders
TO CLASSIFY THE EPILEPTIC PHENOTYPE SEVERITY OF DS PATIENTS | Through study completion, an average of 2 years
  Mild epilepsy will be defined by: i) no history of myoclonic and/or absence seizure, ii) no history of status epilepticus, iii) seizure frequency less than weekly. Patients not fulfilling these criteria will be considered as having severe epilepsy.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy